CLINICAL TRIAL: NCT00441831
Title: The Revolutions of Helicobacter Pylori Infection, Bacterial Density, and Histological Features After Antrectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Mackay Memorial Hospital, secretary, Mackay Memorial Hospital
Other Study IDs: MMH-I-S-261
Record Dates: First submitted 2007-02-27; First posted 2007-03-01 (Estimated); Last update posted 2009-02-05 (Estimated); Status verified 2009-02

CONDITIONS: Helicobacter Pylori Infection; Peptic Ulcer; Bile Reflux; Gastritis
Keywords: Helicobacter pylori infection; peptic ulcer disease; distal partial gastrectomy; bile reflux; gastritis; gastrectomy
MeSH Terms: conditions — Peptic Ulcer; Bile Reflux; Gastritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Helicobacter pylori (HP) is a gram-negative bacillus responsible for one of the most common infections found in humans worldwide. By the early-to-mid 1990s, further evidence emerged supporting the link between the chronic gastritis of HP infection and malignancy in adults, specifically gastric lymphoma and adenocarcinoma. The potential of HP eradication for the prevention of gastric cancer was underlined. At the national consensus meeting held in Brussels in 1998, HP eradication was strongly recommended in past or current peptic ulcer diseases, regardless of activity, complication and post endoscopic resection of early cancer. Some patients received gastric surgery due to the complications of peptic ulcer such as bleeding or perforation in the pre-HP eradication era. Their HP infection status was not surveyed and unknown at the time. Afterward, some of them were not suggested to receive an eradication therapy and recovered from the operative procedure. According to the consensus to treat HP for a purpose to reduce the risk of gastric cancer, these patients were still under risk. There have been only a few surveys on the prevalence of persistent HP infection in patients who have undergone surgery. The aim of the study was to evaluate the prevalence and histological features of HP infection after a time course of partial distal gastric surgery.

DETAILED DESCRIPTION:
The eradication of H pylori is known to reduce the recurrence rate of peptic ulcer and gastric inflammation. But it is still not clear about the prevalence of HP infection in patients after surgical interventions when the micro-environment had been changed. Since biliary enterogastric reflux is suggested to inhibit the growth of HP, we will investigate in a prospective study the effect of partial gastrectomy on the influence of HP infection incidence.

Patients with previous distal gastrectomy will be prospectively evaluated as study group. Same number of patients with the same indication of endoscopy evaluations and without previous gastrectomy will be established as a normal control group for H pylori infection rate comparison. All patients in study and control groups who had previously received H pylori eradication therapy will be excluded. Three gastric biopsy specimens were collected from each patient for histological analysis. Patients with a pre-operative biopsy, operative specimen revealing H pylori colonization or a positive serum H pylori IgG will be indicated previous H pylori infection and will be assessed the percentage of spontaneous clearance of HP infection. A positive bile staining will indicate biliary enterogastric reflux. This assessment will be made by two investigators, and disagreements will be resolved by joint discussion to reach a consensus. Tissue sections stained with hematoxylin and eosin and the Giemsa stain will be examined by pathologist who was unaware of the endoscopy findings. Density of HP in the tissue and histological gastritis activity and intestinal metaplasia will be graded as normal (0), mild (1), moderate (2) and severe (3) based on the Sydney system. Follicular gastritis will be based on the absence (0) or presence (1) of lymphoid follicules and lymphoid with germinal center (2).

The primary end point will be the change of infection rate on HP after distal gastrectomy procedure comparing the normal control. The secondary end point will assess the correlation between the duration of the antrectomy, the operative procedure, the severity of bile reflux with the inhibition of HP growth. Finally, this study will be base on histopathological features with the density of HP, the grading of gastritis activity, intestinal metaplasia and follicular gastritis.

ELIGIBILITY:
Inclusion Criteria:

* Previous distal gastrectomy

Exclusion Criteria:

* Post HP eradication therapy

Ages: 15 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with previous distal gastrectomy
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2007-02; Study Completion 2008-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ming-Jen Chen, M.D.,M.S., Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Division of Gastroenterology, Department of Internal Medicine, Mackay Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Fukuhara K, Osugi H, Takada N, Takemura M, Lee S, Taguchi S, Kaneko M, Tanaka Y, Fujiwara Y, Nishizawa S, Kinoshita H. Duodenogastric reflux eradicates Helicobacter pylori after distal gastrectomy. Hepatogastroenterology. 2004 Sep-Oct;51(59):1548-50. PMID 15362798
- [Background] Huang WH, Wang HH, Wu WW, Lai HC, Hsu CH, Cheng KS. Helicobacter pylori infection in patients with ulcer recurrence after partial gastrectomy. Hepatogastroenterology. 2004 Sep-Oct;51(59):1551-3. PMID 15362799
- [Background] Malfertheiner P, Megraud F, O'Morain C, Bazzoli F, El-Omar E, Graham D, Hunt R, Rokkas T, Vakil N, Kuipers EJ. Current concepts in the management of Helicobacter pylori infection: the Maastricht III Consensus Report. Gut. 2007 Jun;56(6):772-81. doi: 10.1136/gut.2006.101634. Epub 2006 Dec 14. PMID 17170018
- [Background] Johannesson KA, Hammar E, Stael von Holstein C. Mucosal changes in the gastric remnant: long-term effects of bile reflux diversion and Helicobacter pylori infection. Eur J Gastroenterol Hepatol. 2003 Jan;15(1):35-40. doi: 10.1097/00042737-200301000-00007. PMID 12544692